CLINICAL TRIAL: NCT00475319
Title: Late Phase 2 Study of OPC-12759 Ophthalmic Suspension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 037E-06-001
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Results first posted 2013-06-05 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-05

CONDITIONS: Dry Eye Syndromes
Keywords: Dry Eye Syndromes; OPC-12759
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): 0% OPC-12759 ophthalmic suspension received one drop to both eyes four times a day for 4 weeks.
  Interventions: Drug: placebo
- 1% OPC-12759 ophthalmic suspension (Experimental): 1% OPC-12759 ophthalmic suspension received one drop to both eyes four times a day for 4 weeks.
  Interventions: Drug: 1% OPC-12759 ophthalmic suspension
- 2% OPC-12759 ophthalmic suspension (Experimental): 2% OPC-12759 ophthalmic suspension received one drop to both eyes four times a day for 4 weeks.
  Interventions: Drug: 2% OPC-12759 ophthalmic suspension

INTERVENTIONS:
Drug: placebo — comparison of different dosages of drug
  Arms: Placebo
Drug: 1% OPC-12759 ophthalmic suspension — comparison of different dosages of drug
  Arms: 1% OPC-12759 ophthalmic suspension
Drug: 2% OPC-12759 ophthalmic suspension — comparison of different dosages of drug
  Arms: 2% OPC-12759 ophthalmic suspension

SUMMARY:
The purpose of this study is to evaluate the dose-response of OPC-12759 suspension in dry eye patients

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient
2. Subjective complaint of dry eye that has been present for minimum 20 months
3. Ocular discomfort severity is moderate to severe
4. Corneal - conjunctival damage is moderate to severe
5. Unanesthetized Schirmer's test score of 5mm/5minutes or less
6. Best corrected visual acuity of 0.2 or better in both eyes

Exclusion Criteria:

1. Presence of anterior segment disease or disorder other than that associated with keratoconjunctivitis sicca
2. Ocular hypertension patient or glaucoma patient with ophthalmic solution
3. Anticipated use of any topically-instilled ocular medications or patients who cannot discontinue the use during the study
4. Anticipated use of contact lens during the study
5. Patient with punctal plug
6. Any history of ocular surgery within 12 months
7. Female patients who are pregnant, possibly pregnant or breast feeding
8. Known hypersensitivity to any component of the study drug or procedural medications
9. Receipt of any investigational product within 4 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Satoshi Oshima, Study Director — Division of dermatologicals and ophthalmologicals
Locations (6):
- Japan (6):
  - Chubu Region
  - Kansai Region
  - Kanto Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

REFERENCES:
- [Derived] Kinoshita S, Awamura S, Oshiden K, Nakamichi N, Suzuki H, Yokoi N; Rebamipide Ophthalmic Suspension Phase II Study Group. Rebamipide (OPC-12759) in the treatment of dry eye: a randomized, double-masked, multicenter, placebo-controlled phase II study. Ophthalmology. 2012 Dec;119(12):2471-8. doi: 10.1016/j.ophtha.2012.06.052. Epub 2012 Sep 23. PMID 23009892

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in Japan between 2007 and 2008
Pre-assignment Details: Participant flow results are based on the safety set.
Groups:
- 1% OPC-12759 Groups: 1% OPC-12759 ophthalmic suspension received one drop of to both eyes four times a day for 4 weeks
- 2% OPC-12759 Groups: 2% OPC-12759 ophthalmic suspension received one drop of to both eyes four times a day for 4 weeks
- Placebo: 0% OPC-12759 ophthalmic suspension received one drop of to both eyes four times a day for 4 weeks
Period: Overall Study
Arm/Group | 1% OPC-12759 Groups | 2% OPC-12759 Groups | Placebo
Started | 103 | 102 | 103
Completed | 101 | 101 | 99
Not Completed | 2 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% OPC-12759 Groups | 2% OPC-12759 Groups | Placebo | Total
Number analyzed (Participants) | 103 | 102 | 103 | 308
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 70 | 61 | 62 | 193
  >=65 years | 33 | 41 | 41 | 115
Age Continuous [Mean (Standard Deviation); unit: years] | 53.7 (16.6) | 56.3 (16.9) | 55.6 (17.2) | 55.2 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 86 | 90 | 269
  Male | 10 | 16 | 13 | 39
Region of Enrollment [Number; unit: participants]
  Japan | 103 | 102 | 103 | 308

OUTCOME MEASURES:

1. Primary Outcome: Change in Fluorescein Corneal Staining (FCS) Score From Baseline to Last Observation Carried Forward (LOCF)
Description: FCS indicates the damage to the corneal epithelium. Per the National Eye Institute/Industry Workshop report, the cornea was divided into 5 fractions, each of which was given a staining score from 0 to 3, and the total score was calculated(0-15). 0 is better.The change from baseline (CFB) to LOCF at the end of instillation (LOCF endpoint) was used to analyze dose-response. A general linear model was used to examine if slope parameters were not equal to zero.
Time Frame: Baseline, 4weeks
Measure: Mean (Standard Deviation); unit: FCS score
Arm/Group | 1% OPC-12759 Ophthalmic Suspension | 2% OPC-12759 Ophthalmic Suspension | Placebo
Number analyzed (Participants) | 103 | 102 | 103
FCS score | -3.5 (2.2) | -3.7 (2.4) | -1.8 (2.0)
Statistical Analysis 1: Comparison: 1% OPC-12759 Ophthalmic Suspension vs 2% OPC-12759 Ophthalmic Suspension vs Placebo; Test type: Superiority or Other; p = 0.001, t-test, 2 sided — versus placebo; a general linear model

2. Secondary Outcome: Change in Lissamine Green Conjunctival Staining (LGCS) Score From Baseline to Last Observation Carried Forward (LOCF)
Description: LGCS indicates the damage to the conjunctival epithelium. Per the National Eye Institute/Industry Workshop report, the conjunctival sac and the conjunctina was divided into 6 ractions, each of which was given a staining score from 0 to 3, and the total score was calculated(0-18). 0 is better. The CFB to each study time point was compared between the active-drug groups and the placebo group, and LOCF endpoint scores were used to compare the active-drug groups and the placebo group. In each treatment group, baseline scores and those obtained at each study time point were compared.
Time Frame: Baseline, 4weeks
Measure: Mean (Standard Deviation); unit: LGCS score
Arm/Group | 1% OPC-12759 Groups | 2% OPC-12759 Groups | Placebo
Number analyzed (Participants) | 103 | 102 | 103
LGCS score | -4.0 (2.8) | -4.5 (2.9) | -1.9 (3.0)
Statistical Analysis 1: Comparison: 1% OPC-12759 Groups vs 2% OPC-12759 Groups vs Placebo; Test type: Superiority or Other; p = 0.001, t-test, 2 sided — versus placebo; a general linear model

ADVERSE EVENTS:
Arm/Group | 1% OPC-12759 Groups | 2% OPC-12759 Groups | Placebo
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/102 | 1/103
Other Adverse Events (participants affected / at risk) | 30/103 | 31/102 | 27/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1% OPC-12759 Groups (N=103) | 2% OPC-12759 Groups (N=102) | Placebo (N=103)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1% OPC-12759 Groups (N=103) | 2% OPC-12759 Groups (N=102) | Placebo (N=103)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 2 (2) | 1 (1) | 2 (2)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Corneal erosion (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 4 (4) | 2 (2) | 5 (5)
Iritis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Eyelids pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 3 (3) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood potassium increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Glucose urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 14 (14) | 16 (16) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No